CLINICAL TRIAL: NCT00218660
Title: Naltrexone and Psychosocial Treatments for the Treatment of Cocaine Dependence Complicated by Alcohol Dependence
Brief Title: Naltrexone in Two Models of Psychosocial Treatments for Cocaine and Alcohol Dependence - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-5186-1; P60DA005186 (NIH); P60-5186-1
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2010-06

CONDITIONS: Alcoholism; Cocaine Dependence
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Nal + BRENDA
  Interventions: Drug: Naltrexone; Behavioral: BRENDA
- 2 (Placebo Comparator): Placebo + BRENDA
  Interventions: Behavioral: BRENDA; Drug: Placebo
- 3 (Experimental): Nal + CBT
  Interventions: Drug: Naltrexone; Behavioral: CBT
- 4 (Placebo Comparator): Placebo + CBT
  Interventions: Behavioral: CBT; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 150mg/day Naltrexone
  Arms: 1; 3
Behavioral: BRENDA — Psychosocial Treatment
  Arms: 1; 2
Behavioral: CBT — Cognitive Behavioral Therapy
  Arms: 3; 4
Drug: Placebo
  Other Names: 150mg/day Placebo
  Arms: 2; 4

SUMMARY:
The purpose of this study is to see whether naltrexone is safe and useful in preventing alcohol relapse, as well as in decreasing craving for alcohol in people with a diagnosis of alcohol and cocaine dependence. Naltrexone is approved by the Food and Drug Administration (FDA) for the treatment of alcohol dependence. However, the medication was not approved as yet at the dosage we will use in this study. The dosage we will use for the study (150 mg), is greater than the recommended dosage from the Physician's Desk Reference (50mg). Unlike other medicines (like Antabuse) useful in the treatment of alcohol dependence, naltrexone will not make you sick if you drink alcohol. Rather, people who are taking this medication have reported that it helps decrease the pleasure associated with drinking for them. This study is being conducted because the medication (Naltrexone) has not been well studied in people with both alcohol and cocaine dependence, so it is still investigational.

We believe that if we can reduce alcohol consumption through naltrexone and psychotherapy, this may lead to reduced cocaine use. We are also conducting this study to test two different types of psychotherapy as a method for reducing cocaine and alcohol use. One type of psychotherapy, CBT, is designed to help people learn to cope with situations that put them at high risk for relapse to cocaine and/or alcohol use. The other type of psychotherapy, BRENDA, will use focuses on strengthening motivation to recover from cocaine and/or alcohol use, and on developing techniques to handle possible barriers to recovery. We seek to enroll 300 patients in the study.

DETAILED DESCRIPTION:
The project will use a 2x2 design to assess the efficacy of naltrexone for treating subjects who are both cocaine and alcohol dependent and who will receive either CBT or BRENDA alone or in combination with naltrexone. There will be 300 DSM-IV cocaine-alcohol dependent male and female subjects randomized to one of four groups (75 subjects per group). Subjects will be randomized to either 150mg/day naltrexone or placebo and to receive either CBT (a type of cognitive behavior therapy derived from relapse prevention principles), or a new primary-care basedmodel, BRENDA, comprised of strategies for enhancing motivation and treatment compliance. All subjects will receive one of the four combinations of medication and psychosocial treatment. The length of the study for each subject includes one week of screening/baseline assessments, 12 weeks of double-blind, placebo-controlled naltrexone treatment combined with one of two psychosocial treatments, and a 6-month and 12-month follow-up visit. Following successful completion of detoxification (abstinence from alcohol and cocaine for 7 days), informed consent will be signed, and Week 1 will be devoted to completing screening and baseline measures. In Week 2, subjects will be randomly assigned to medication/ psychosocial treatment combination. Following completion of the 12-week, double-blind treatment trial, subjects will be evaluated at 6-month and 12-months post-treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, 18-65 years old.
* Meets DSM-IV criteria for current diagnoses of cocaine and alcohol dependence, determined by the SCID.
* In the past 30 days, S used no less than $200-worth of cocaine and >15 standard alcohol drinks (avg)/week with at least 1 day of 4 or more drinks, determined by the TLFB--adapted to collect daily cocaine use.
* Successful completion of alcohol detoxification, i.e.,
* 5 consecutive days of abstinence from cocaine and alcohol, via self-reports and negative urine toxicology screens.
* Lives a commutable distance to the TRC and agrees to follow-up visits.
* Understands and signs the consent.

Exclusion Criteria:

* Abstinent from cocaine or alcohol for 30 days prior to signing consent form. (S may have been institutionalized in the prior month and still be eligible if his/her cocaine and alcohol use that month met inclusion criteria.)
* Current DSM-IV diagnosis of any substance dependence other than cocaine, alcohol, nicotine, or cannabis determined by the SCID.
* Evidence of opiate use in the past 30 days, determined by self-report on the SCID or ASI, and/or by a urine drug screen that is positive for opiates at treatment entry.
* Current treatment with psychotropic medications (excluding short-term use of benzodiazepines for detoxification), including disulfiram.
* History of unstable or serious medical illness, including need for opioid analgesics.
* History of epilepsy or seizure disorder.
* Known severe physical or medical illnesses such as AIDS, active hepatitis, significant hepatocellular injury as evidenced by elevated bilirubin levels, or elevated levels over 4.5x normal of aspartate aminotransferase (AST), and serum glutamic-pyruvic transaminase (SGPT).
* Current severe psychiatric symptoms, e.g., psychosis, dementia, acute suicidal or homicidal ideation, mania or depression requiring antidepressant therapy, or which would make it unsafe for the patient to participate in the opinion of the primary investigators.
* Use of an investigational medication in the past 30 days.
* Female Ss who are pregnant, nursing, or not using a reliable method of contraception. [Note: Criteria 4-10 will be assessed via the medical exam plus results from lab tests.]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 1998-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Alcohol and Cocaine use during the treatment trial period and at the 6- and 12-month follow-up. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Pettinati HM, Kampman KM, Lynch KG, Suh JJ, Dackis CA, Oslin DW, O'Brien CP. Gender differences with high-dose naltrexone in patients with co-occurring cocaine and alcohol dependence. J Subst Abuse Treat. 2008 Jun;34(4):378-90. doi: 10.1016/j.jsat.2007.05.011. Epub 2007 Jul 30. PMID 17664051
- [Derived] Ueland GA, Dahl SR, Methlie P, Hessen S, Husebye ES, Thorsby PM. Adrenal steroid profiling as a diagnostic tool to differentiate polycystic ovary syndrome from nonclassic congenital adrenal hyperplasia: pinpointing easy screening possibilities and normal cutoff levels using liquid chromatography tandem mass spectrometry. Fertil Steril. 2022 Aug;118(2):384-391. doi: 10.1016/j.fertnstert.2022.05.012. Epub 2022 Jun 18. PMID 35725670
- [Derived] Ueland GA, Methlie P, Oksnes M, Thordarson HB, Sagen J, Kellmann R, Mellgren G, Raeder M, Dahlqvist P, Dahl SR, Thorsby PM, Lovas K, Husebye ES. The Short Cosyntropin Test Revisited: New Normal Reference Range Using LC-MS/MS. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1696-1703. doi: 10.1210/jc.2017-02602. PMID 29452421